CLINICAL TRIAL: NCT06015490
Title: The Impact of the Physiological Response to Sugar on Brain Activity and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Alexandra DiFeliceantonio, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: #23-297
Record Dates: First submitted 2023-05-03; First posted 2023-08-29 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Food Preferences; Appetitive Behavior
MeSH Terms: conditions — Food Preferences; Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sucrose, then Glucose, then Fructose (Experimental): Participants will consume a 110 kcal sucrose drink 6 times during 1 week. Then, they will consume a 110 kcal glucose drink 6 times during 1 week, and then, a 110 kcal fructose drink 6 times during 1 week.
  Interventions: Other: Sucrose drink; Other: Glucose drink; Other: Fructose drink
- Sucrose, then Fructose, then Glucose (Experimental): Participants will consume a 110 kcal sucrose drink 6 times during 1 week. Then, they will consume a 110 kcal fructose drink 6 times during 1 week, and then, a 110 kcal glucose drink 6 times during 1 week.
  Interventions: Other: Sucrose drink; Other: Glucose drink; Other: Fructose drink
- Glucose, then Fructose, then Sucrose (Experimental): Participants will consume a 110 kcal glucose drink 6 times during 1 week. Then, they will consume a 110 kcal fructose drink 6 times during 1 week, and then, a 110 kcal sucrose drink 6 times during 1 week.
  Interventions: Other: Sucrose drink; Other: Glucose drink; Other: Fructose drink
- Glucose, then Sucrose, then Fructose (Experimental): Participants will consume a 110 kcal glucose drink 6 times during 1 week. Then, they will consume a 110 kcal sucrose drink 6 times during 1 week, and then, a 110 kcal fructose drink 6 times during 1 week.
  Interventions: Other: Sucrose drink; Other: Glucose drink; Other: Fructose drink
- Fructose, then Glucose, then Sucrose (Experimental): Participants will consume a 110 kcal fructose drink 6 times during 1 week. Then, they will consume a 110 kcal glucose drink 6 times during 1 week, and then, a 110 kcal sucrose drink 6 times during 1 week.
  Interventions: Other: Sucrose drink; Other: Glucose drink; Other: Fructose drink
- Fructose, then Sucrose, then Glucose (Experimental): Participants will consume a 110 kcal fructose drink 6 times during 1 week. Then, they will consume a 110 kcal sucrose drink 6 times during 1 week, and then, a 110 kcal glucose drink 6 times during 1 week.
  Interventions: Other: Sucrose drink; Other: Glucose drink; Other: Fructose drink

INTERVENTIONS:
Other: Sucrose drink — Participants will consume flavored beverage solutions containing 110 calories of sucrose in 6 exposure sessions within 1 week. One exposure session will include pre- and post-consumption blood draws and indirect calorimetry measurements inside a metabolic chamber over a 2-hour period. The other 5 exposure sessions will occur at specified times outside the laboratory sessions. Subjective ratings of internal state (i.e., hunger, fullness, and thirst) will be collected throughout each exposure. Subjective ratings of liking and wanting of each beverage will also be assessed.
  Other Names: Flavored beverage solution with 110 calories of sucrose
Other: Glucose drink — Participants will consume flavored beverage solutions containing 110 calories of glucose in 6 exposure sessions within 1 week. One exposure session will include pre- and post-consumption blood draws and indirect calorimetry measurements inside a metabolic chamber over a 2-hour period. The other 5 exposure sessions will occur at specified times outside the laboratory sessions. Subjective ratings of internal state (i.e., hunger, fullness, and thirst) will be collected throughout each exposure. Subjective ratings of liking and wanting of each beverage will also be assessed.
  Other Names: Flavored beverage solution with 110 calories of glucose
Other: Fructose drink — Participants will consume flavored beverage solutions containing 110 calories of fructose in 6 exposure sessions within 1 week. One exposure session will include pre- and post-consumption blood draws and indirect calorimetry measurements inside a metabolic chamber over a 2-hour period. The other 5 exposure sessions will occur at specified times outside the laboratory sessions. Subjective ratings of internal state (i.e., hunger, fullness, and thirst) will be collected throughout each exposure. Subjective ratings of liking and wanting of each beverage will also be assessed.
  Other Names: Flavored beverage solution with 110 calories of fructose

SUMMARY:
The goal of this pilot study is to test the feasibility of assessing how biological factors and chemical properties of sugars may influence metabolism and food reward in humans. The main questions it aims to answer are:

• Can differences in appetitive responses and neural activations to sucrose (table sugar) and its chemical components (glucose and fructose) be measured and quantified?

This study is a crossover design, meaning every participant will complete every condition. Participants will consume beverages containing sucrose, glucose, or fructose, which are each novelly flavored, 6 times within a week. During one of the consumption times, energy expenditure, carbohydrate oxidation, and blood glucose will be measured in the lab before and for 2 hours after consumption. After participants have consumed each condition, they will undergo a tasting task in the MRI scanner, neural responses to receipt of the beverages are measured.

DETAILED DESCRIPTION:
Prior studies in humans indicate that while energy expenditure response is similar after consumption of equal amounts of fructose, glucose, and sucrose (a dimer of glucose + fructose), carbohydrate oxidation and blood glucose responses differ. Elevated carbohydrate oxidation responses appear to be driven by the presence of fructose, and elevated blood glucose responses appear to be driven by the presence of glucose. Prior work also suggests that post-ingestive signals of glucose availability, measure specifically as blood glucose levels, intestinal glucose transporter activity, and carbohydrate oxidation rate, are all associated with elevated brain response to calorie-predictive flavor cues and reward learning of these flavor cues. However, in animal models, glucose has been shown to repeatedly and reliably condition these calorie-predictive learning responses, but fructose does not. Human work has indicated that oxidation of glucose is critical for these responses. Thus, it is unclear what roles fructose and glucose each play in conditioning reward responses and flavor-calorie learning. We hypothesize that fructose plays a synergistic role in enhancing flavor-calorie learning without itself conditioning the reward response.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 18.5-25 kg/m2
2. Not pregnant or planning to become pregnant during study participation
3. Residing in the Roanoke area and/or willing/able to attend sessions at the Fralin Biomedical Research Institute (FBRI) at Virginia Tech Carilion
4. Weigh at least 110 lbs

Exclusion Criteria:

1. Current inhaled nicotine use
2. History of alcohol dependence.
3. Current or past diagnosis of cardiometabolic disease or problems, including diabetes, endocrine, heart, or thyroid problems, that may influence study outcomes
4. Hemoglobin A1C >5.7%
5. Taking medications known to influence study measures (including attention-deficit/hyperactivity disorder (ADHD), allergy, antidepressant, antipsychotic, anxiolytic, birth control, blood pressure, blood glucose, cholesterol, thyroid, sleep, or weight loss medications)
6. Active medical or neurologic disorder, including cardiometabolic conditions or gastrointestinal conditions that may influence study outcomes
7. Recent change in body weight (gain or loss of > 5 lbs within the past 3 months)
8. Current shift work (typical pattern of work/activity overnight)
9. Previous weight loss surgery
10. Adherence to a special diet within the past 3 months (e.g., low-carb or ketogenic diet, exclusion of food groups/specific macronutrients, intermittent fasting, etc.)
11. Allergy to any food or ingredient included in the study diets, meals, or beverages
12. Currently pregnant or planning to become pregnant during study participation
13. Claustrophobia
14. Contraindications for MRI, including pacemaker, aneurysm clips, neurostimulators, cochlear or other implants, metal in eyes, regular work with steel, etc. (Note: This is an fMRI-specific exclusion criterion. Participants may be allowed to participate in all other study sessions and measures that do not involve fMRI.)
15. Contraindications for bioelectrical impedance analysis, specifically implanted devices
16. Use of substances (or combinations of substances) in doses and frequencies that could influence neural outcomes of study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at Virginia Tech Carilion, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First CS Intervention (1 Week)
Arm/Group | Sucrose, Then Glucose, Then Fructose | Sucrose, Then Fructose, Then Glucose | Glucose, Then Fructose, Then Sucrose | Glucose, Then Sucrose, Then Fructose | Fructose, Then Glucose, Then Sucrose | Fructose, Then Sucrose, Then Glucose
Started | 1 | 2 | 0 | 1 | 1 | 2
Completed | 1 | 2 | 0 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second CS Intervention (1 Week)
Arm/Group | Sucrose, Then Glucose, Then Fructose | Sucrose, Then Fructose, Then Glucose | Glucose, Then Fructose, Then Sucrose | Glucose, Then Sucrose, Then Fructose | Fructose, Then Glucose, Then Sucrose | Fructose, Then Sucrose, Then Glucose
Started | 1 | 2 | 0 | 1 | 1 | 2
Completed | 1 | 2 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Period: Third CS Intervention (1 Week)
Arm/Group | Sucrose, Then Glucose, Then Fructose | Sucrose, Then Fructose, Then Glucose | Glucose, Then Fructose, Then Sucrose | Glucose, Then Sucrose, Then Fructose | Fructose, Then Glucose, Then Sucrose | Fructose, Then Sucrose, Then Glucose
Started | 1 | 2 | 0 | 1 | 1 | 1
Completed | 1 | 2 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to the glucose, then fructose, then sucrose arm/order
Groups:
- Total: Total of all reporting groups
Arm/Group | Sucrose, Then Glucose, Then Fructose | Sucrose, Then Fructose, Then Glucose | Glucose, Then Fructose, Then Sucrose | Glucose, Then Sucrose, Then Fructose | Fructose, Then Glucose, Then Sucrose | Fructose, Then Sucrose, Then Glucose | Total
Number analyzed (Participants) | 1 | 2 | 0 | 1 | 1 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (0) | 28.5 (0.7) |  | 42 (0) | 31 (0) | 22 (1.4) | 28.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 |  | 0 | 0 | 1 | 2
  Male | 1 | 1 |  | 1 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 |  | 1 | 1 | 2 | 7
  Unknown or Not Reported | 0 | 0 |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0 | 0 | 0
  Asian | 1 | 1 |  | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 |  | 1 | 0 | 0 | 1
  White | 0 | 1 |  | 0 | 1 | 2 | 4
  More than one race | 0 | 0 |  | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 |  | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 |  | 1 | 1 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Preference- Subjective Liking Ratings for Each Beverage on a Scale
Description: Subjective ratings of liking of flavors used in the intervention will be assessed at baseline and after the intervention. The generalized Labeled Magnitude Scale will be used. The scale is anchored by descriptors of "Most Disliked Sensation Imaginable" and "Most Liked Sensation Imaginable" at the lower and upper ends, respectively. The score is determined by the place on the scale participants select (range of scale is 0-100). An increase in score from baseline to post-intervention indicates an increase in liking.
Time Frame: Immediately after informed consent and in the post-test session approximately 5 weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Glucose Drink; Fructose Drink; Sucrose Drink: Participants complete behavioral preference tests for conditions at baseline and after the conditioning paradigm in a post-test. All participants complete all conditions in a cross-over design.
Arm/Group | Glucose Drink | Fructose Drink | Sucrose Drink
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | -12.8 (26.3) | -12.0 (26.2) | -12.6 (26.3)

2. Secondary Outcome: Post-Test Measure of Preference- Subjective Wanting Ratings for Each Beverage on a Scale
Description: Subjective ratings of liking of flavors used in the intervention will be assessed at baseline and after the intervention. A Visual Analog Scale will be used. Participants select a place on the line that corresponds with their subjective rating, and the score is determined by the place selected (range of scores is 0-100). The line is anchored by polar opposite descriptors ("Do not want at all" and "Want very much"). An increase in score from baseline to post-intervention indicates and increase in wanting.
Time Frame: At the end of study; approximately 5 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glucose Drink | Sucrose Drink | Fructose Drink
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 42 (12.7) | 54.8 (12.5) | 46.9 (14.5)

3. Secondary Outcome: Post-Test Measure of Preference - Wanting (ad Libitum Intake): The Amount Consumed of Each Beverage is Reported as the Outcome
Description: Ad libitum intake will be used as a measure of wanting in a post-test session. Participants will be provided each beverage used during the intervention and asked to drink as much or as little of them as they would like over a 30-minute period.
Time Frame: At the end of study; approximately 5 weeks after first session
Measure: Mean (Standard Deviation); unit: ml consumed
Arm/Group | Glucose Drink | Fructose Drink | Sucrose Drink
Number analyzed (Participants) | 6 | 6 | 6
ml consumed | 67.8 (98.1) | 66.0 (99.1) | 66.3 (98.5)

4. Secondary Outcome: Post-Test Measure of Preference- Wanting (Forced Choice): Number of Participants Who Chose Each Indicated Beverage
Description: Forced choice will be used as a measure of wanting in a post-test session. Participants will be provided each of the beverages used during the intervention and asked to choose 1 to take home with them.
Time Frame: At the end of study; approximately 5 weeks after first session
Population: In the post-test session, participants are asked to choose among the Glucose, Sucrose, and Fructose Drinks which they would like to take home in a forced choice test. Participants are only allowed to choose one of the three conditions.
Measure: Count of Participants; unit: Participants
Arm/Group | Glucose Drink | Fructose Drink | Sucrose Drink
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 3 | 2

5. Secondary Outcome: Blood Oxygen Level-dependent (BOLD) Response to Beverages
Description: In a post-test session, functional magnetic resonance imaging (fMRI) scans were performed while beverages (without calories) used during the intervention and a tasteless solution are delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids. Participants receive the glucose, sucrose, fructose, and tasteless (control) solutions 18 times each over the course of 2 runs. Contrasts of interest are the blood oxygen level-dependent (BOLD) response of glucose+>tasteless solution, sucrose>tasteless solution, and fructose>tasteless deliveries. Parameter estimates for these contrasts are extracted and reported. A positive outcome reflects greater whole-brain BOLD response for the sugar condition compared with a tasteless solution.
Time Frame: At the end of study; approximately 5 weeks after first session
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Glucose Drink: In a post-test, beverages (without calories) used during the intervention were delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids during functional magnetic resonance imaging (fMRI). Outcomes presented here are blood oxygen-level dependent (BOLD) response for the contrast of glucose>tasteless solution delivery.
- Fructose Drink: In a post-test, beverages (without calories) used during the intervention were delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids during functional magnetic resonance imaging (fMRI). Outcomes presented here are blood oxygen-level dependent (BOLD) response for the contrast of fructose>tasteless solution delivery.
- Sucrose Drink: In a post-test, beverages (without calories) used during the intervention were delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids during functional magnetic resonance imaging (fMRI). Outcomes presented here are blood oxygen-level dependent (BOLD) response for the contrast of sucrose>tasteless solution delivery.
Arm/Group | Glucose Drink | Fructose Drink | Sucrose Drink
Number analyzed (Participants) | 6 | 6 | 6
arbitrary units | 0.005 (0.085) | 0.109 (0.186) | 0.050 (0.210)

6. Secondary Outcome: Blood Glucose Response to Beverages
Description: Blood glucose will be assessed at baseline and at set time points for 2 hours after consumption of intervention beverages (baseline, 5-, 20-, 40-, 60-, 90-, and 120-minutes after drink consumption)in one exposure session. Area under the curve is calculated using these time points and reported as the outcome measure.
Time Frame: Each week for 3 weeks during the study
Population: One participant withdrew from the study prior to the glucose and sucrose drink sessions but completed the fructose drink session.
Measure: Mean (Standard Deviation); unit: mg/dl*min
Groups:
- Glucose Drink; Fructose Drink; Sucrose Drink: Blood draws occur before and at 6 time points after consumption of a research study drink during a lab session. Blood glucose is assessed and area under the curve for blood glucose is calculated.
Arm/Group | Glucose Drink | Fructose Drink | Sucrose Drink
Number analyzed (Participants) | 6 | 7 | 6
mg/dl*min | 16821.25 (4861.348755) | 11484.58334 (1468.61789) | 13760.66666 (3813.485448)

7. Secondary Outcome: Energy Expenditure in Response to Beverages
Description: Indirect calorimetry will be used to determine energy expenditure at baseline and for 120 minutes after consumption of condition beverages in an exposure session. Area under the curve is calculated as a change from baseline energy expenditure using minute-by-minute resolution across 120 minutes and reported as the outcome measure.
Time Frame: Each week for 3 weeks during the study
Population: Technical challenges with equipment and data collection resulted in lower sample size for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: kcal/min*min
Groups:
- Glucose Drink; Fructose Drink; Sucrose Drink: Energy expenditure is assessed with indirect calorimetry before and for 2 hours after consumption of a research study drink during a lab session. Area under the curve for energy expenditure is calculated.
Arm/Group | Glucose Drink | Fructose Drink | Sucrose Drink
Number analyzed (Participants) | 5 | 6 | 6
kcal/min*min | -0.89 (6.63) | 0.940 (6.14) | 1.89 (3.86)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: No participants were randomized to the glucose drink first, then fructose drink, then sucrose drink arm/order.
Groups:
- Sucrose Drink: Participants will consume a 110 kcal sucrose drink 6 times during 1 week.
- Fructose Drink: Participants will consume a 110 kcal fructose drink 6 times during 1 week.
- Glucose Drink: Participants will consume a 110 kcal glucose drink 6 times during 1 week.
Arm/Group | Sucrose Drink | Fructose Drink | Glucose Drink
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT06015490/Prot_SAP_000.pdf